CLINICAL TRIAL: NCT02768428
Title: Effectiveness of Knowledge by Video and Handbook to Measure Knowledge of Liver Cancer Patients With First Trans-arterial Chemoembolization (TACE)
Brief Title: Effectiveness of Knowledge by Video and Handbook of Liver Cancer Patients With First Trans-arterial Chemoembolization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulabhorn Hospital (Other)
Responsible Party: Principal Investigator, Ruechuta Molek, Registered Nurse, Chulabhorn Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 017/2015
Record Dates: First submitted 2016-04-18; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
Keywords: Knowledge [K01.468]; Video-Audio Media [V01.255.500]; Handbooks [V02.520]
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video-Audio Media (Experimental): watching the entire video in 15 mins
  Interventions: Other: Video-Audio Media
- Handbooks (No Intervention): study the hand book in 15 mins

INTERVENTIONS:
Other: Video-Audio Media — each arm spends 15 mins for watching the video or study the handbooks
  Other Names: Handbooks
  Arms: Video-Audio Media

SUMMARY:
Objective: To compare the effectiveness between Video and Handbook on providing knowledge of TACE.

Study Design: A prospective, randomized, controlled trial.

DETAILED DESCRIPTION:
Background : Liver cancer is a serious disease with a high death rate. One of the treatment modalities for liver cancer is TACE. Patients always scare of the first TACE due to their lack of knowledge and inadequate comprehension of the procedure. Hence, they crave to have a good quality in nursing service. Researcher would like to compare the effectiveness knowledge between Video and Handbook regarding patients' health education.

Objective: To compare the effectiveness between Video and Handbook on providing knowledge of TACE.

Study Design: A prospective, randomized, controlled trial.

Setting: Chulabhorn Hospital, Bangkok, THAILAND.

Methods : Eighty liver cancer patients are included in the study. They are systematically computerized and randomized into two groups - an experiment or video group (N 40) and a control or Handbook group (N = 40). A 40-item exam is performed to test the patients' knowledge before (x score), after (y score) and 60 days (z score) after the procedure. The 15-min study was taken in an isolated room. The points of interest are the effectiveness of medias on learning achievement and relative growth of knowledge. The relative growth of knowledge (G1, G2 score) was calculated as follows:

G1 = 100 (Y-X)/(F-X) % ; G2 = 100 (Z-X)/(F-X)%

Retention of knowledge (R) = 100 - (G1 - G2) %

Where G = Relative growth of knowledge R = Retention of knowledge X = Pre-test score Y = Post-test score Z = Final-test score F = Total score

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 75 years
* Willing to participate the study
* 1st TACE
* Can comprehend all information in video or handbook
* No trouble of hearing
* Can complete the 40-item test

Exclusion Criteria:

* Have psychological/mental problems

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
knowledge about TACE (A 40-item exam is performed to test the patients' knowledge) | 2 years
  The points of interest are the effectiveness of medias on learning achievement and relative growth of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Ruechuta Molek, MNS, Principal Investigator — Chulabhorn Hospital
Locations (1):
- Chulabhorn Hospital, Thailand, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Varela M, Real MI, Burrel M, Forner A, Sala M, Brunet M, Ayuso C, Castells L, Montana X, Llovet JM, Bruix J. Chemoembolization of hepatocellular carcinoma with drug eluting beads: efficacy and doxorubicin pharmacokinetics. J Hepatol. 2007 Mar;46(3):474-81. doi: 10.1016/j.jhep.2006.10.020. Epub 2006 Nov 29. PMID 17239480
- [Background] McCurdy HM. Improving outcomes for patients receiving transarterial chemoembolization for hepatocellular carcinoma. Gastroenterol Nurs. 2013 Mar-Apr;36(2):114-20. doi: 10.1097/SGA.0b013e318288c8be. PMID 23549214
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Result] Soerjomataram I, Lortet-Tieulent J, Parkin DM, Ferlay J, Mathers C, Forman D, Bray F. Global burden of cancer in 2008: a systematic analysis of disability-adjusted life-years in 12 world regions. Lancet. 2012 Nov 24;380(9856):1840-50. doi: 10.1016/S0140-6736(12)60919-2. Epub 2012 Oct 16. PMID 23079588